CLINICAL TRIAL: NCT04580485
Title: A Phase 1, Open-Label, Multicenter Study of INCB106385 as Monotherapy or in Combination With Immunotherapy in Participants With Advanced Solid Tumors
Brief Title: INCB106385 Alone or in Combination With Immunotherapy in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 106385-102; 2020-002921-27 (EudraCT Number)
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Bladder Cancer; Non Small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Cancer; Castration Resistant Prostate Cancer; Colorectal Cancer; Gastric/ Gastroesophageal Junction; Hepatocellular Carcinoma; Pancreatic Ductal Adenocarcinoma; Squamous Carcinoma of the Anal Canal
Keywords: INCB106385; Advanced Solid Tumors; PD-1
MeSH Terms: conditions — Ovarian Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Masking Description: Open Label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (TGA) - INCB106385 (Experimental): In part 1 dose escalation, the dose levels will be escalated following a BOIN design.
  In part 2 dose expansion, participants will be assigned to different groups based on their tumor types and treated at the RDE.
  Interventions: Drug: INCB106385
- Treatment Group B (TGB) - INCB106385+INCMGA00012 (Experimental): In part 1 dose escalation, the dose levels will be escalated following a BOIN design.
  In part 2 dose expansion, participants will be assigned to different groups based on their tumor types and treated at the RDE.
  Interventions: Drug: INCB106385; Drug: INCMGA00012

INTERVENTIONS:
Drug: INCB106385 — INCB106385 will be administered orally QD
Drug: INCMGA00012 — INCMGA0012 will be administered IV once every 4 weeks (Q4W)
  Arms: Treatment Group B (TGB) - INCB106385+INCMGA00012

SUMMARY:
This is a multicenter, open-label, dose-escalation/dose-expansion Phase 1 clinical study to investigate the safety, tolerability, PK profile, pharmacodynamics, and preliminary clinical efficacy of INCB106385 when given as monotherapy or in combination with INCMGA00012 in participants with selected CD8 T-cell-positive advanced solid tumors including SCCHN, NSCLC, ovarian cancer, CRPC, TNBC, bladder cancer, and specified GI malignancies (defined as CRC, gastric/GEJ cancer, HCC, PDAC, or SCAC)

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign an ICF.
* Willing and able to conform to and comply with all Protocol requirements.
* Histologically or cytologically confirmed advanced/metastatic SCCHN, NSCLC, ovarian cancer, TNBC, CRPC, bladder cancer, and specified GI malignancies (defined as CRC, gastric/GEJ cancer, HCC, PDAC, or SCAC) that progressed after treatment with available therapies (including anti PD-(L)1 therapy (if applicable).
* Willingness to undergo pre- and on-treatment tumor biopsy.
* Have CD8 T-cell-positive tumors.
* Presence of measurable disease according to RECIST v1.1.
* ECOG performance status 0 to 1.
* Life expectancy > 12 weeks.
* Willingness to avoid pregnancy or fathering children based.
* Acceptable laboratory parameters

Exclusion Criteria:

* Clinically significant cardiac disease.
* Known or active CNS metastases and/or carcinomatous meningitis.
* Active or inactive autoimmune disease or syndrome that required systemic treatment in the past 2 years or receiving systemic therapy for an autoimmune or inflammatory disease..
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses > 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment.
* Known additional malignancy that is progressing or requires active treatment,or history of other malignancy within 2 years of the first dose of study treatment.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study treatment.
* Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis.
* Immune-related toxicity during prior immune therapy for which permanent discontinuation of therapy is recommended, or any immune-related toxicity requiring intensive or prolonged immunosuppression to manage.
* Any prior chemotherapy, biological therapy, or targeted therapy to treat the participant's disease within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Any prior radiation therapy within 28 days before the first dose of study treatment.
* Undergoing treatment with another investigational medication or having been treated with an investigational medication within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Concomitant treatment with strong CYP3A4 inhibitors or inducers.
* Receipt of a live vaccine within 30 days of the first dose of study treatment.
* Infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week of the first dose of study treatment.
* Evidence of HBV or HCV infection or risk of reactivation.
* Known history of HIV (HIV 1/2 antibodies).
* History of organ transplant, including allogeneic stem-cell transplantation.
* Known hypersensitivity or severe reaction to any component of study drug(s) or formulation components.
* Presence of a gastrointestinal condition that may affect drug absorption.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study,pose a significant risk to the participant; or interfere with interpretation of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAE) | Up to Approximately 28 months
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 90 days after last dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCB106385 as a single agent or in combination with INCMGA00012 | Up to 6 months
  Maximum observed plasma concentration.
Tmax of INCB106385 as a single agent or in combination with INCMGA00012 | Up to 6 months
  Time to maximum plasma concentration
Cmin of INCB106385 as a single agent or in combination with INCMGA00012 | Up to 6 months
  Minimum observed plasma concentration over the dose interval
AUC of INCB106385 as a single agent or in combination with INCMGA00012 | Up to 6 months
  Area under the plasma concentration-time curve
CL/F of INCB106385 as a single agent or in combination with INCMGA00012 | Up to 6 months
  Apparent oral dose clearance
Objective Response Rate (ORR) | Up to approximately 24 months
  Defined as the percentage of participants with a best overall response of CR or PR, as determined by investigator radiographic disease assessment according to RECIST v1.1.
Disease Control Rate | Up to approximately 24 months
  Defined as the percentage of participants with a best overall response of CR, PR, or SD, as determined by investigator radiographic disease assessment according to RECIST v1.1.
Duration Of Response (DOR) | Up to approximately 24 months
  Defined as the time from the earliest date of CR or PR until the earliest date of disease progression, as determined by investigator radiographic disease assessment according to RECIST v1.1, or death due to any cause if occurring sooner than progression.
Change in tumoral gene expression | Predose and Week 5-6
  Defined as the percent of patients with change in tumoral targeted gene expression compared to baseline
Change in immune cell activation in tumors | Predose and Week 5-6
  Defined as the percent of patients demonstrating change in immune cell activation in tumors compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Rybicka, M.D, Study Director — Incyte Corporation
Locations (27):
- United States (8):
  - Cedars-Sinai Medical Center, West Hollywood, California
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Belgium (2):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- France (3):
  - Institut Bergonie, Bordeaux
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - A.O.U. Di Modena - Policlinico, Modena
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona
- Spain (5):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Clinica Universidad de Navarra (Cun), Pamplona
- United Kingdom (5):
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - University of Glasgow, Glasgow
  - Guys and St Thomas Nhs Foundation Trust, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - The Christie Nhs Foundation Trust Uk, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency